CLINICAL TRIAL: NCT07407686
Title: Improving the Engagement of Underserved Communities With the Prostate Cancer Genetics Service: Identifying Barriers & Facilitators and Developing Supportive Resources Using a Co-production and Collaborative Approach
Brief Title: Improving Engagement From Underserved Communities With Prostate Cancer Genetics Services
Acronym: INCLUDE PC
Status: Not yet recruiting | Type: Observational
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 361063
Record Dates: First submitted 2025-11-21; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Prostate Cancer
Keywords: qualitative research methods; co-production; MRC Complex Intervention Developement; Health Literacy and Health Behaviour Theories; Prostate cancer screening in high risk groups; semi-structured interviews and focus groups; reflexive thematic analysis of qualitative data; Evaluation of outputs
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Surveys and Questionnaires; Focus Groups

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Semi-structured interview participants: Up to 60 participants for semi-structured interviews, 20 from each of the following underserved groups in prostate cancer screening; Black African and Black Caribbean, transgender and non-binary with a prostate, reduced access to healthcare.
  Interventions: Other: Surveys; Other: Semi-structured interviews and focus groups

INTERVENTIONS:
Other: Surveys — Up to 30 surveys with 10 of these individuals undergoing short interviews to assess the improvement of their understanding around prostate cancer
Other: Semi-structured interviews and focus groups — Up to 60 total semi-structured interviews (up to 20 per underserved group) to assess barriers and facilitators to prostate cancer screening and how they would like information to improve their understanding to be presented.

SUMMARY:
Earlier work explored barriers and facilitators to accessing prostate cancer screening, particularly in underserved communities, and provided valuable insights to build upon.

This study will explore perspectives on how genetic risk for prostate cancer is explained and understood through in-depth interviews with members of underserved communities. Findings from this work, alongside earlier results, will be used to co-design clear and accessible digital educational resources in collaboration with community members and relevant charities.

Participation in cancer screening programmes in the UK varies, with differences linked to socioeconomic status, ethnicity and health literacy. Similar inequalities are seen in access to prostate cancer genetics services, indicating a need for improved engagement.

Successful integration of genetics into prostate cancer care requires clear and inclusive information about genetic testing processes, possible outcomes and interpretation of results. Currently, there are limited resources explaining genetic risk for prostate cancer in an accessible way.

Co-production with representatives from underserved communities will ensure that educational materials are understandable, relevant and acceptable to all.

DETAILED DESCRIPTION:
There is variability in uptake of cancer screening programmes in the UK with participation affected by socioeconomic status, ethnicity & health literacy. This lack of representation is also seen within the prostate cancer genetics service, suggesting that further work is required to promote engagement. The successful mainstream integration of genetics into prostate cancer management will require people to understand the process, potential outcomes and interpretation of results. In addition, the information provided should be inclusive.

The barriers and facilitators to accessing prostate cancer screening work commenced under a service evaluation (CCR SE1284). This project provided valuable data from underserved communities which we wish to build on. This study aims to further explore perspectives on genetic risk explanation and education in further depth using semi-structured interviews and to use these and earlier findings to co-design educational digital materials to raise awareness about prostate cancer and genetic risk measurement, in keeping with the wishes from the communities that have worked with us.

Development of educational multi-media materials:

Utilising the Medical Research Council's Complex Intervention Design Framework, we will co-design educational materials, using the data collected from community champions and relevant charities.

Evaluation of educational multi-media materials:

The co-designed education materials will undergo evaluation in a pilot phase and then again after dissemination. Methods of evaluation will be adopted to include acceptability, usability and integration into clinical practice.

There are few current resources explaining the genetic risk of prostate cancer and opportunities to participate in genetic risk studies. The study will work alongside representatives from underserved communities to ensure that educational materials developed are accessible and acceptable to all.

ELIGIBILITY:
Inclusion Criteria:

1. Men and people with prostates age 18 and above
2. Those who belong to the three underserved groups; Black African and Black Caribbean Ancestry, transgender and non-binary people with a prostate and those with reduced access to healthcare
3. We allow intersectionality within reason and will narratively describe any instances of these in the writeup of findings
4. Those who are able to freely consent to inclusion
5. Individuals with and without a lived experience of prostate cancer

Exclusion Criteria:

1. To avoid exhaustion, we will only allow participation in two interview or focus groups per individual for the entirety of the study
2. Those without capacity to consent to interview (capacity is assumed unless there is good reason to believe otherwise)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men and people with prostates from the following three communities:
  * Black African and Black Caribbean
  * Transgender women and non-binary people with prostates
  * Reduced access to healthcare
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-02-28 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of educational materials, demonstrating that users have an increase in understanding or prostate cancer risk and symptoms as well as genetic risk. | February 2026 to August 2026
  Using surveys (before and after use of resources) and interviews to measure improvement in understanding in individuals without experience of prostate cancer.
Increased representation from underserved groups in the referrals to our genetic research studies. | As soon as the educational materials are live, which we aim to be from June 2026, increase in referrals to our genetic research studies from under-represented groups will be measured. This will take place for 12 months.
  Using demographic data from referrals via our website to our genetic research studies
Qualitative data such as hits to the webpage and scroll depth and how many have signed up to the genetic research studies via the website. | These data will be collected from as soon as the webpage goes live for the subsequent 12 months.
  This is a short term measure of how effective and engaging the resources are.

SECONDARY OUTCOMES:
Improved representation of underrepresented groups in our genetic risk studies. | Measurements of the demographics of our research participants takes place currently. Any signficant change in representation will be reported for a minimum 12 months after the webpage and resources go live.
  Recruits to our genetic research studies will be screened for demographics.
Reduced barriers to prostate cancer screening and participation in genetic research faced by underrepresented communities | The web page will go live in July 2026 and will be a long term resource (many years), regularly updated by our team. There will also be rounds of evaluation, using surveys and interviews, with subsequent adaption.
  These resources will be distributed by the community champions who we have co-designed them with. These community champions have social media networks with a strong following in their respective community and they are trusted by community members. Therefore, the resources and the webpage will have a far reach within the community to encourage engagement with empowering information and to promote prostate cancer screening and participation with our genetic risk studies.

CONTACTS AND LOCATIONS:
Overall Officials: Ros Eeles, Study Chair — Institute of Cancer Research, United Kingdom

IPD SHARING:
Plan to Share IPD: No
There will be no confidential data shared outside of the research team and the study participants are members of the public, not patients.